CLINICAL TRIAL: NCT06565572
Title: An Open-label Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for PCARP (Posterior Column Ataxia with Retinitis Pigmentosa) Disease Due to Mutations in FLVCR1
Brief Title: Antisense Oligonucleotide Treatment for PCARP Disease Due to Mutation in FLVCR1
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-2313
Record Dates: First submitted 2023-08-09; First posted 2024-08-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-08

CONDITIONS: Posterior Column Ataxia with Retinitis Pigmentosa
MeSH Terms: conditions — Posterior column ataxia with retinitis pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- nL-FLVC-001 Arm (Experimental): nL-FLVC-001 is an antisense oligonucleotide that will be injected into the vitreous
  Interventions: Drug: nL-FLVC-001

INTERVENTIONS:
Drug: nL-FLVC-001 — nL-FLVC-001 is an antisense oligonucleotide that will be injected into the vitreous

SUMMARY:
The goal of this clinical trial is to evaluate a specific antisense oligonucleotide medication in one patient with posterior column ataxia with retinitis pigmentosa. The main question it aims to answer is: what is the safety and tolerability of this medication in a single participant.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s).
* Genetically confirmed FLVCR1-related disease.
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.

Exclusion Criteria:

* Allergy to any of the ASO components
* Participant has any condition that in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Over 12 months
We will measure visual acuity, retinal thickness, examine changes in fundus photos and biomicroscopic exam post nL-FLVC-001 administration in a participant with FLVCR1 gene mutation | Over 12 months

SECONDARY OUTCOMES:
Measure any changes in the Cardiff Visual Ability Questionnaire for Children (CVAQC-25) in one patient with PCARP after nL-FLVC-001 intravitreal injection. | Over 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States